CLINICAL TRIAL: NCT04459533
Title: The Use of Neuromuscular Blockade Monitor as a Strategy for Neuromuscular Blockade Agents Saving in ICU COVID-19 Patients
Brief Title: Sparing in Neuromuscular Blockade in COVID 19 ICU
Acronym: TOF-COVID
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 2020_TOF-COVID
Record Dates: First submitted 2020-06-22; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Neuromuscular Blockade; Human Characteristics; Complication of Medical Care; Intensive Care Unit Acquired Weakness
Keywords: neuromuscular blockade agent; neuromuscular blockade monitor; Train of Four (TOF); critical illness; COVID 19
MeSH Terms: conditions — Critical Illness; COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TOF group: COVID-19 patients admitted to the ICU, receiving mechanical ventilation and NMB agents, for whom a NMB monitor use (TOF) was reported in the electronic health records (EHR).
  Interventions: Device: TOF protocol
- Control group: COVID-19 patients admitted to the ICU, receiving mechanical ventilation and NMB agents, with no NMB monitor use reported in the EHR

INTERVENTIONS:
Device: TOF protocol — To the introduction of CISATRACURIUM, Initial bolus was at 0.2mg/kg and initial continuous infusion at 0.18mg/kg/h of theoretical ideal weight.
  To the introduction of ATRACURIUM, initial bolus was at 0.5mg/kg and initial continuous infusion at 0.5mg/kg/h of theoretical ideal weight.
  Introduction of NMBA was associated to deep sedation (RASS - 4 or RAMSAY 6; BIS 40 to 60).
  TOF was measured through the electric stimulation of peripheral nerves (facial or ulnar nerve).
  The dose of NMB agents was then adapted according to the number of answers to the TOF, per 4 hours:
  * If 0 response and no respiratory asynchrony: no change in flow rate
  * If >=1 or respiratory asynchrony: increase of the continuous curare flow by 20% preceded by a bolus identical to the one administered at the beginning of NMB agent, then recheck at H+1.
  Groups: TOF group

SUMMARY:
This is a retrospective case-controlled study of the effect of the use of a neuromuscular blockade (NMB) monitor on the consumption of NMB agents in patients under mechanical ventilation in the context of COVID-19.

The use of NMB agents during mechanical ventilation in patients with acute respiratory distress syndrome (ARDS) improves respiratory support conditions and reduces mortality. In the context of COVID-19 pandemic, patients with severe forms of the disease hospitalized in intensive care units (ICU) benefit from prolonged mechanical ventilation with frequent use of NMB agents. Large amount of such patient admitted in a short time has led to a shortage of NMB agents, particularly cisatracurium.

The use of NMB monitors (for example - Train of Four (TOF)) is a well-established practice in general anesthesia. There is no recommendation for the use of NMB monitor in ICU patients available up to date. However, in the attempt to reduce the consumption of NMB agents a NMB monitoring was used in ICU patients during the COVID-19 pandemic at university hospitals of Hospices Civil de Lyon, with the endorsement of the local College of Anesthetists.

The aim of our study is to evaluate if the use of a NMB monitor decreases the consumption of NMB agents in patients under mechanical ventilation in the context of COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* PCR-proven SARS-CoV-2 infection
* Use of VM (mechanical ventilation)
* Use of NMB agents for at least 48 hours

Exclusion Criteria:

* Pregnancy
* extracorporeal membrane oxygenation (ECMO)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We included all COVID patients in ICU university hospitals in Lyon who required mechanical ventilation and NMB for at least 48 hours.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
NMB agents consumption | ICU discharge an average of 4 weeks
  We measured the total NMB agents consumption during the stay: cisatracurium and/or atracurium (milligram). Nurses report continuous infusion rates of NMB agents. By extracting this data we were able to retrieve the total approximate dose (we're missing the bolus doses).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine, Hôpital de la Croix Rousse, Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: No